CLINICAL TRIAL: NCT00604331
Title: Effects of Pyruvate in Patients With Cardiogenic Shock and Intra-aortic Balloon Counterpulsation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herzzentrum Goettingen (Other)
Responsible Party: Gerd Hasenfuss/Professor Dr. med., Cardiology and Pneumology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PYR-2008-01; 12/10/00
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Shock, Cardiogenic; Heart Failure; Acute Myocardial Infarction
Keywords: Pyruvic Acid; Shock, Cardiogenic; Catecholamines; Intra-Aortic Balloon Pumping; Cardiac Output; Cardiac Index; Cardiac Function
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure | interventions — Pyruvic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator): Pyruvate
  Interventions: Drug: Pyruvate

INTERVENTIONS:
Drug: Pyruvate — sodium pyruvate 300 mmol/L, 360 mL/h i.c. over 30 minutes.

SUMMARY:
Pyruvate is an intermediate of energy metabolism and was shown to possess pronounced positive inotropic effects in vitro and in vivo without altering myocardial oxygen consumption. Moreover, it was shown that the effects of beta-adrenergic stimulation were potentiated. Thus, it might be possible to save catecholamines in patients with severe heart failure or cardiogenic shock. This study was designed to test the hemodynamic effects of pyruvate administered into a coronary artery in addition to intra-aortic balloon pump counterpulsation in patients with severe heart failure or in patients with acute myocardial infarction and cardiogenic shock after having performed percutaneous coronary intervention. A pronounced improvement in hemodynamics is expected to occur.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients male/female
* Age: 18 - 85 years
* Weight: 45 - 110 kg
* Height 150 - 195 cm
* Clinically signs of heart failure (NYHA III-IV) refractary to therapy or cardiogenic shock in acute myocardial infarction
* written informed consent or witnessed verbal consent or presumed will (compassionate use)

Exclusion Criteria:

* Malignoma
* Clinically significant cardiac valve stenosis
* Participation in another clinical trial with relevant or probable drug-interactions
* Pregnancy or lactation
* Addiction
* Poor compliance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | 60 minutes

SECONDARY OUTCOMES:
Cardiac Index | 60 minutes
Arterial Pressure | 60 minutes
Pulmonary capillary wedge pressure | 60 minutes
Pulmonary artery pressure | 60 minutes
systemic vascular resistance | 60 minutes
pulmonary vascular resistance | 60 minutes
heart rate | 60 minutes
stroke volume | 60 minutes
catecholamine need | 60 minutes
safety | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Hasenfuss, Prof. Dr., Principal Investigator — Herzzentrum Goettingen, Cardiology and Pneumology
Locations (1):
- Herzzentrum Goettingen, Cardiology and Pneumology, Göttingen, Germany

REFERENCES:
- [Background] Hermann HP, Pieske B, Schwarzmuller E, Keul J, Just H, Hasenfuss G. Haemodynamic effects of intracoronary pyruvate in patients with congestive heart failure: an open study. Lancet. 1999 Apr 17;353(9161):1321-3. doi: 10.1016/s0140-6736(98)06423-x. PMID 10218531
- [Result] Schillinger W, Hunlich M, Sossalla S, Hermann HP, Hasenfuss G. Intracoronary pyruvate in cardiogenic shock as an adjunctive therapy to catecholamines and intra-aortic balloon pump shows beneficial effects on hemodynamics. Clin Res Cardiol. 2011 May;100(5):433-8. doi: 10.1007/s00392-010-0261-4. Epub 2010 Dec 4. PMID 21132310